CLINICAL TRIAL: NCT03834701
Title: Safety and Efficacy of Endoscopic Ultrasound-guided RadioFrequency Ablation for the Treatment of Functional and Non-functional Pancreatic NeuroEndocrine Neoplasms: A Multicenter Prospective Study
Brief Title: Endoscopic Ultrasound-guided RadioFrequency Ablation for the Treatment Pancreatic NeuroEndocrine Neoplasms
Acronym: RAPNEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPNEN
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Carcinoma; Pancreas Neoplasm; Neuroendocrine Tumor Gastrointestinal, Hormone-Secreting
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS guided radiofrequency ablation (Experimental): Radiofrequency ablation will be performed using a system that consists of an 19-gauge needle electrode (140-cm long), a radiofrequency generator, and an inner cooling system that circulates chilled saline solution during the RFA procedure.
  Interventions: Device: EUS guided radiofrequency ablation

INTERVENTIONS:
Device: EUS guided radiofrequency ablation — The EUS-RFA system (Taewoong, Seoul, Korea) utilized for EUS-RFA consists of an 19-gauge needle electrode (140-cm long), a radiofrequency generator, and an inner cooling system that circulates chilled saline solution during the RFA procedure. The inner metal part is insulated over its entire length, with the exception of the terminal 5 to 20mm for energy delivery. The needle electrode is attached to a radio frequency current generator (VIVA RF generator; Taewoong) and to a cooling pump. The generator, in addition to providing radio frequency current, allows the control of physical power and impedance parameters.

SUMMARY:
This study evaluates the possibility and the safety of performing local therapy for Pancreatic neuroendocrine neoplasms (PanNENs) using radiofrequency ablation of the tumor under ultrasonography (EUS) guidance.

DETAILED DESCRIPTION:
Pancreatic neuroendocrine neoplasms (PanNENs) are rare, but their incidence has significantly increased in the last decades. The mainstay treatment of PanNENs is surgery, which is associated with a significant benefit in term of survival but also with significant short- and long-term adverse events.

Based on the above data, less invasive alternative therapeutic interventions to avoid short- and long-term adverse events of surgery are needed.

In this context radiofrequency ablation has been reported to be effective in the treatment of these tumors in absence of major adverse events. However, the available studies on the matter are limited by small sample size and lack of standardized criteria for patient selection.

ELIGIBILITY:
Inclusion Criteria:

For all patients

* Age ≥18 years and <80 years
* Signed written informed consent
* Distance from the main pancreatic duct ≥2mm
* Able to undergo endoscopic ultrasound examination
* Homogeneous enhancement at contrast harmonic EUS (CH-EUS)

For patients with functional pancreatic neuroendocrine neoplasms (F-PanNENs), almost all insulinomas

* Definitive diagnosis of a clinical syndrome related to excessive insulin secretion fasting test, insulin blood levels, C-peptide blood levels)
* Single lesion visualized at CT, and/or MRI, and/or EUS
* Size < 20mm

For patients with non functional pancreatic neuroendocrine neoplasms (NF-PanNENs)

* EUS fine needle biopsy (FNB) proven NF-PanNENs
* 68Ga-DOTATATE PET/CT positive for a pancreatic lesion and negative for lymph nodes, liver, and other distant metastases
* Hyper- or Iso-enhancing pattern at MRI and/or CT with negative lymph nodes, liver, and other distant metastases
* G1 or G2 ≤ 5% on histological examination of EUS-guided biopsy samples utilizing EUS-FNB needles
* Diameter between 15mm and 25mm,
* Absence of symptoms
* Absence of inner calcifications

Exclusion Criteria:

* For all patients
* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma (FFP)
* Use of anticoagulants that cannot be discontinued
* INR >1.5 or platelet count <50.000
* Previous inclusion in other studies
* Pregnancy
* Minimal distance from the main pancreatic duct <1mm
* Inability to sign the informed consent
* Heterogeneous enhancement at contrast harmonic EUS (CH-EUS)

For patients with F-PanNENs (almost all insulinomas)

* Diagnosis work up negative excessive hormone secretion syndrome
* Multiple lesions visualized at CT, and/or MRI, and/or EUS
* Size > 20mm
* For patients with NF-PanNENs
* G2>5% or G3 on histological examination of EUS-guided biopsy samples
* Diameter <15 mm and >25 mm
* Presence of symptoms
* Presence of calcifications
* Hypo-enhancing pattern at MRI and/or CT
* 68Ga-DOTATATE PET/CT positive for lymph nodes, liver, and other distant metastasis
* Diagnosis on multiple endocrine neoplasia type 1 (MEN1) syndrome or Von Hippel Lindau syndrome
* Previous inclusion in other studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) after EUS-guided radiofrequency ablation (RFA) | 1 year
  AEs will be classified as procedural when they occur during the procedure; post-procedural when they will occur up to 14 days after the procedure; late when they will occur more than 14 days after the procedure. Minor AEs will be those that need no therapy and have no sequelae (A) or have minor therapy or consequence, including overnight admission (B). Major events include those that require major therapy or hospitalization (24- 48 hours) (C); major therapy, need unplanned increase in level of care, or hospitalization >48 hours (D); or result in permanent adverse sequelae (E) and death (F).

SECONDARY OUTCOMES:
Rates of secondary surgery | 1 year
  Number of patients who will require secondary surgey due to adverse events occurence, no response/failed or partial/recurrence outcome to the RFA treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Larghi, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma, RM
  - Universita' del Sacro Cuore, Rome

REFERENCES:
- [Derived] Hofland J, de Herder WW, Kann PH. Turning Up the Heat: Endoscopic Ablation of Pancreatic Neuroendocrine Neoplasms. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5053-5055. doi: 10.1210/jc.2019-00954. No abstract available. PMID 31058975